CLINICAL TRIAL: NCT01622621
Title: Randomized Phase II Trial of Stereotactic Body Radiotherapy (SBRT) Versus Sublobar Resection for High-Risk Patients With Early Stage Non-Small Lung Cancer (NSCLC)
Brief Title: Stereotactic Body Radiotherapy (SBRT) Versus Sublobar Resection for High-Risk Patients Non-Small Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Unable to enroll to the randomized arm.
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Dennis Wigle, MD, PhD, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11-000805
Record Dates: First submitted 2012-06-15; First posted 2012-06-19 (Estimated); Last update posted 2020-09-11 (Actual); Status verified 2020-09

CONDITIONS: Lung Neoplasms
Keywords: Lung; Cancer
MeSH Terms: conditions — Lung Neoplasms; Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Randomized Sublobar Resection (Active Comparator): Randomized by computer to receive a sublobar resection.
  Interventions: Procedure: Sublobar Resection
- Randomized SBRT (Active Comparator): Randomized by computer to receive Stereotactic Body Radiotherapy (SBRT).
  Interventions: Radiation: Stereotactic Body Radiotherapy (SBRT)
- Observation Sublobar Resection (Active Comparator): Patient decides with doctor to undergo a sublobar resection.
  Interventions: Procedure: Sublobar Resection
- Observation SBRT (Active Comparator): Patient decides with doctor to undergo SBRT.
  Interventions: Radiation: Stereotactic Body Radiotherapy (SBRT)

INTERVENTIONS:
Procedure: Sublobar Resection — Undergo surgery which removes a sublobar resection of the lung
  Arms: Observation Sublobar Resection; Randomized Sublobar Resection
Radiation: Stereotactic Body Radiotherapy (SBRT) — 54 Gy in 3 fractions
  Arms: Observation SBRT; Randomized SBRT

SUMMARY:
This randomized phase II trial is for medically inoperable early stage non-small cell lung cancer (NSCLC) patients. It is designed to compare the number of patients who are disease free and alive at 2 years between Stereotactic Body Radiotherapy (SBRT) and surgical intervention arms. SBRT is less invasive and felt to be equally effective to surgery for early stage NSCLC. Surgery is currently the standard of care for these patients. The hypothesis of this study is that SBRT is at least as good as surgery for disease free survival at 2 years.

DETAILED DESCRIPTION:
The current standard of care for Stage I Non-Small Lung Cancer (NSCLC) is sublobar surgical resection. Recent trials have suggested that early stage NSCLC might be successfully treated with SBRT amongst those who are medically inoperable. SBRT is the precise delivery of a high dose of radiation to control tumors while limiting damage to surrounding normal tissues. Patients on the SBRT arm will receive 54 Grays (Gy) in 3 fractions. One gray is the absorption of one joule of energy, in the form of ionizing radiation, per kilogram of matter. Recent advances with three-dimensional conformal and Intensity Modulated Radiotherapy (IMRT) techniques can now compensate for lung motion and allow delivery of high-dose, single fractions to the primary lung tumor for patients with clinical state I NSCLC.

Local control and survival results appear promising. SBRT for early stage lung cancer may offer a potentially equivalent, non-invasive treatment alternative to surgical resection. Additionally, SBRT may be associated with fewer complications and better quality of life. SBRT may be an acceptable or even preferred treatment option in higher-risk patients not able to tolerate a surgical lobectomy. This clinical dilemma is increasingly faced in our lung cancer practice at Mayo Clinic, with no comparative effectiveness data to guide treatment decisions.

Patients will be evaluated by both Thoracic Surgery and Radiation Oncology. Randomization can occur through either group but a patient must see both in consultation prior to randomization. For patients meeting enrollment criteria but unwilling to participate in randomization, observational arms for each of SBRT and sublobar resection will enroll up to 24 patients as part of the 96 patient total.

The patients will receive the following tests as part of their clinical care:

* Computed Tomography (CT)-Positron Emission Tomography (PET) will be used for mediastinal imaging
* Endobronchial/endoscopic ultrasound (EBUS/EUS)-Fine Needle Aspiration (FNA) or mediastinoscopy will be used for pathologic assessment of level 2 lymph nodes (N2) greater than 1 cm in the short axis on CT scan and/or SUV greater than 1.5 fold background
* Follow-up CT scans at 6 months, 12 months, 18 months, and 24 months for the Surgery and SBRT groups.
* Follow-up Pulmonary Function Tests at 1 year

ELIGIBILITY:
Inclusion Criteria

* Patients must have a suspicious lung nodule for clinical stage I NSCLC.
* Pathologic confirmation at the time of surgery is acceptable. Patients randomized to SBRT require core biopsy for diagnosis prior to treatment.
* Patient must have a mass ≤ 5 cm maximum diameter by CT size estimate that is clinical stage I (T1N0, T2N0)
* Patient must have a CT scan of the chest and upper abdomen and PET-scan within 60 days prior to date of registration.
* Patient must have an Eastern Cooperative Oncology Group (ECOG) or Zubrod performance status 0, 1, or 2.
* Patient must meet at least one major criteria or meet a minimum of two minor criteria as described below:

Major Criteria:

* Forced expiratory volume in one second (FEV1) ≤ 50% predicted
* Carbon monoxide diffusing capacity (DLCO) ≤ 50% predicted

Minor Criteria:

* Age ≥75
* FEV1 51-60% predicted
* DLCO 51-60% predicted
* Pulmonary hypertension (defined as a pulmonary artery systolic pressure greater than 40 mmHg) as estimated by echocardiography or right heart catheterization
* Poor left ventricular function (defined as an ejection fraction of 40% or less)
* Resting or Exercise Arterial oxygen partial pressure (pO2) ≤ 55 mm Hg or blood oxygen saturation (SpO2) ≤ 88%
* pCO2 > 45 mm Hg
* Modified Medical Research Council (MMRC) Dyspnea Scale ≥ 3.

Exclusion Criteria

* Patient must not have had previous intra-thoracic radiation therapy.
* No prior malignancy except adequately treated non-melanoma skin cancer, in situ cervical cancer, localized prostate cancer, stage 0 Chronic lymphocytic leukemia (CLL), or other cancer disease-free > 3 yrs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-05; Primary Completion 2017-04-25 (Actual); Study Completion 2017-04-25 (Actual)

PRIMARY OUTCOMES:
Number of patients alive at 2 years (Overall Survival [OS]) | 2 years after treatment
  All patients who are alive at 2 years.

SECONDARY OUTCOMES:
Number of patients with disease free survival (DFS) at 2 years | 2 years after treatment
  All patients who are alive and free of disease at 2 years. Disease burden will be determined by computed tomography.

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Wigle, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States